CLINICAL TRIAL: NCT00287625
Title: To Study the Effect of Early Pulmonary Rehabilitation on Exacerbations, Hospitalization Rates and Quality of Life in Patients Admitted to Hospital With Acute Exacerbation of Chronic Obstructive Pulmonary Disease.
Brief Title: Early Pulmonary Rehabilitation for Hospitalized Patients With Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr. Fanny WS Ko, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resp/ko/2006/001
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- 1 (Active Comparator): PRP
  Interventions: Procedure: Pulmonary rehabilitation
- 2 (No Intervention): control

INTERVENTIONS:
Procedure: Pulmonary rehabilitation — Pulmonary rehabilitation
  Arms: 1

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a disease state characterized by airflow limitation that is not fully reversible. Acute exacerbation of COPD (AECOPD) with increasing symptoms like dyspnea, cough and sputum is the natural history of the disease and incurs significant burden to our health care system. In Hong Kong, COPD was the 5th leading cause of death, and accounted for at least 4% of all public hospital acute admissions in 2003. Previous studies have shown that pulmonary function and quality of life were adversely affected by frequent exacerbations. Strategies to decrease the heavy use of health care resources is urgently needed for the benefits of the patients and the society.

Pulmonary rehabilitation programme (PRP) is a multidisciplinary programme of care for patients with chronic respiratory impairment. In COPD patients, the programme can be tailored individually and can optimize each patient's physical and social performance and autonomy. Previous studies on patients with stable COPD found that a PRP including education and physical training could lead to statistically significant and clinically meaningful improvements in health related quality of life and exercise capacity.

COPD patients who just have experienced an episode of acute exacerbations are at high risk of developing another attack. There has been only one randomized controlled study looking at the effect of out-patient PRP for patients immediately after an exacerbation. It has shown that PRP immediately after an exacerbation was safe and improved the exercise capacity and the quality of life at 3 months. However, the follow up duration of the study was short and thus the effect of rehabilitation on recurrent exacerbations and hospitalizations is not assessed and this information is important.

The investigators would thus like perform a randomized controlled trial to assess if a short course (for 6 weeks) out-patient PRP for patients admitted to acute hospital for AECOPD could have a positive impact on the patients by decreasing their health care resources utilization (recurrent COPD exacerbations, hospitalizations and accident and emergency department [AED] attendance) and improving the quality of life of the patients over a period of 1 year. Patients will be randomized to either a control group or PRP intervention group.

It is hope that the information generated from this study will be able to give a guide to whether short course PRP is effective for the patient (in terms of quality of life) and the health care system (in terms of health care utilization).

DETAILED DESCRIPTION:
Patients admitted with AECOPD will be recruited for the study. AECOPD will be defined when a patient with background COPD has at least two of the major symptoms (increased dyspnoea, increased sputum purulence, increased sputum amount) or one major and one minor symptom (nasal discharge/congestion, wheeze, sore throat, cough) for at least two consecutive days.5,17 Inclusion criteria include patients who are ambulatory (no major joint problem and no Class III or IV angina), patients agree to join exercise programme if offered, the forced expiratory volume in 1 second (FEV1) <70% predicted normal and an age of over 40 years old. Patients who have had PRP within the past 1 year will not be recruited for this study.

The subjects will be randomized to 2 groups:

1. Usual care group (Control)
2. PRP group

A random number generator will be used to assign whether the patient is to be in the control or PRP group. The computer programme will help to randomize subjects in equal opportunity in either group but taking into account 5 factors: age (< 70 years or ≥ 70 years),sex, length of hospital admission (< 7 days or ≥ 7 days), 6 minute walk test ( < 100 metres or ≥ 100 metres), and predicted FEV1 (< 30% or ≥ 30%). This method is adapted by the study of Man et al.

After recruitment in the AECOPD admission, baseline assessment will be done 24 hours before discharge from hospital. Each subject will then be followed up every 3 months after discharge for 1 year. For the intervention group, the PRP will start within 10 days of discharge from the hospital. Patients in the intervention group will attend the rehabilitation unit in our physiotherapy department on 3 half days per week for 6 weeks. In the first visit, the patient will be seen by a nurse specialist and offered smoking cessation counseling and inhaler technique will be reinforced. The nurse will also offer psychosocial support to the patient. The exercise sessions will be performed by 2 dedicated physiotherapists. Supervised exercise training includes use of treadmill, arm cycling, and arm and leg weight training will be provided with intensity adjusted by the physiotherapist based on the tolerability and physiological variables (oxygen saturation and heart rate) of the patient. Patients will also be advised to perform home exercises. The physiotherapist will also teach the patient on proper breathing techniques and how to cope with the daily activities.

For the control group, the patients will also be seen by the nurse specialist within 10 days of discharge from the hospital as in the PRP group. The patients will be offered smoking cessation advice and inhaler technique will be reinforced as in the PRP group. Both the control and PRP groups will be followed up every 3 months in our respiratory research clinic. The Standard medications (including inhaled corticosteroid if appropriate according to the GOLD guideline1) will be prescribed to the patients for management of COPD in both groups. Both the PRP group and control group will also be seen by nurse specialist in each visit for further education of the disease and counseling.

Assessments will be performed to monitor the patient's progress in both groups:

1. Lung function test (pre and post bronchodilator) (baseline, 3 month, 6 month, 9 month and 12 month)
2. 6 min walk test (baseline, 3 month, 6 month, 9 month and 12 month)
3. Body mass index measurement (baseline, 3 month, 6 month, 9 month and 12 month)
4. Modified Medical Research Council dyspnoea scale (MMRC)(baseline, 3 month, 6 month, 9 month and 12 month)
5. St George's Respiratory Questionnaire (SGRQ), medical outcomes short form 36 questionnaire (SF-36) and chronic respiratory questionnaire(baseline, 3 months, 12 months)

Exacerbations (that required treatment with a course of oral steroid or antibiotics), AED department visits and hospitalization will be counted. Patient will be phone contacted to check for any mortality if the patient does not return for follow up.

Each patient will be asked to give informed consent and ethical committee approval will be obtained from the Joint The Chinese University of Hong Kong - New Territories East Cluster Clinical Research Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with AECOPD will be recruited for the study. AECOPD will be defined when a patient with background COPD has at least two of the major symptoms (increased dyspnoea, increased sputum purulence, increased sputum amount) or one major and one minor symptom (nasal discharge/congestion, wheeze, sore throat, cough) for at least two consecutive days.
* Inclusion criteria include patients who are ambulatory (no major joint problem and no Class III or IV angina),
* patients agree to join exercise programme if offered, the forced expiratory volume in 1 second (FEV1) <70% predicted normal and an age of over 40 years old.

Exclusion Criteria:

* Patients who have had PRP within the past 1 year will not be recruited for this study.
* Patient who are unable or refuse to consent for the study will also be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Baseline, 3 months, 6 months, 9 months and 12 months

SECONDARY OUTCOMES:
Lung function | Baseline, 3 month, 6 month, 9 month and 12 month
Dyspnoea score | Baseline, 3 month, 6 month, 9 month and 12 month
6 minute walk distance | Baseline, 3 month, 6 month, 9 month and 12 month
Frequency of COPD exacerbation | Baseline, 3 month, 6 month, 9 month and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Fanny WS Ko, MBChB, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Shatin, N.t., Hong Kong